CLINICAL TRIAL: NCT05398900
Title: Validity and Reliability of Indonesian Translated Ages and Stages Questionnaires - Third Edition (ASQ-3) as a Screening Tool for Developmental Delay in 1-12 Months Old Children
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Prof. Hartono Gunardi, MD, PhD, Professor, Indonesia University
Other Study IDs: 0519/UN2.F1/ETIK/PPM.00.02
Record Dates: First submitted 2022-05-25; First posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Developmental Delay; Child Development; Child Development Disorder; Global Developmental Delay; Infant Development; Motor Delay; Speech Delay; Communication Disorders; Development Delay
Keywords: Developmental delay; developmental screening; Indonesian ASQ-3 questionnaire; validity; reliability
MeSH Terms: conditions — Learning Disabilities; Developmental Disabilities; Psychomotor Disorders; Language Development Disorders; Communication Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aimed to provide the validity and reliability of the Indonesian ASQ-3 questionnaires as a screening tool for developmentally delayed children aged less than one year old. This study was divided into 2 phases. The first phase (April-June 2018) included the transcultural adaptation of the ASQ-3 questionnaires for 2 to 12 months age groups from English to Indonesian. The second phase (July- September 2018) included a cross-sectional study of Indonesian ASQ-3 questionnaires for parents/caregivers of children aged 1-12 months, with 35 children in each age group by cluster sampling methods, in 2 district areas in East Jakarta.

ELIGIBILITY:
Inclusion Criteria:

* Parents with children aged 1-12 months
* Parents who finished at least elementary school

Exclusion Criteria:

* Parents with communication difficulties
* Parents who could not speak Indonesian language

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Parents with children aged 1-12 months living in East Jakarta
Sampling Method: Probability Sample
Enrollment: 245 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Child development | 1 day (Once)
  Measured once with Indonesian Ages and Stages-3 questionnaire (cross sectional study) with maximum score of 60 per domain.

CONTACTS AND LOCATIONS:
Locations (1):
- Kampung Melayu subdistrict and Cipinang Muara subdistrict, Jatinegara district, Jakarta, Indonesia